CLINICAL TRIAL: NCT05631444
Title: Comparison of the Therapeutic Potential of Autologous Bone Marrow Mononuclear Cells Versus Allogenic Wharton Jelly-derived Mesenchymal Stem Cells in Diabetic Patients With Chronic Limb-threatening Ischemia
Brief Title: Bone Marrow Mononuclear Cells vs Mesenchymal Stem Cells in Diabetic Patients With Chronic Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Responsible Party: Principal Investigator, Martha Ligia Arango Rodríguez, Director Technical and Scientific Centro de Terapias Avanzadas Fundación Ofalmológica de Santander (FOSCAL), Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLTI 01
Record Dates: First submitted 2022-10-30; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Chronic Limb-threatening Ischemia; Diabetes Mellitus
Keywords: Bone marrow mononuclear cells; Mesenchymal stem cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetes Mellitus | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo group (n=10), which consisted of 15 injections of 1 mL of vehicle (1 mL saline solution with 2% of autologous serum) on periadventitial arteries in one dose at day 0.
  Interventions: Biological: Cell-based therapy
- Auto-BM-MNC (Experimental): Auto-BM-MNC (n=7) were obtained from diabetic patients. Fifteen injections of 7.197x106 ± 2.984x106 cells/mL each with 2% of autologous serum were periadventitial arteries administrated in one dose at day 0.
  Interventions: Biological: Cell-based therapy
- Allo-WJ-MSCs (Experimental): Allo-WJ-MSCs (n=7) were obtained from culturing the WJ from healthy cordon umbilical donors unrelated to the patient. Fifteen injections of 1.333x106 cells/mL each with 5% of human serum albumin serum were periadventitial arteries administrated in one dose at day 0.
  Interventions: Biological: Cell-based therapy

INTERVENTIONS:
Biological: Cell-based therapy — One dose of auto-BM-MNC, one dose of allo-WJ-MSCs, or one dose of placebo solution (saline solution with 2% of autologous serum), were periadventitial arteries administration in CTLI patients.

SUMMARY:
Patients in the severe stages of Chronic limb-threatening ischemia (CLTI) are prone to amputation and death, leading to poor quality of life and a great socioeconomic burden.

There is an urgent need to develop an effective therapeutic strategy to treat this disease. In this context, autologous bone marrow mononuclear cells (BM-MNC) and allogeneic mesenchymal stem cells derived from different sources have emerged as promising therapeutic approaches for this condition.

DETAILED DESCRIPTION:
Comparison of the therapeutic potential of BM-MNC vs. allogeneic Wharton jelly-derived mesenchymal stem cells (allo-WJ-MSCs) in diabetic patients with CLTI.

Twenty-four type 2 diabetic patients in the most severe stages of the CLTI (category 4 or 5 in Rutherford's classification and transcutaneous oxygen pressure (TcPO2) below 30 mm Hg were enrolled and randomized to receive 15 injections of (i) BM-MNC (7.197x106 ± 2.984 x106 cells/mL each with 2% of autologous serum) (n=7), (ii) allo-WJ-MSCs (1.333 x106 cells/mL each with 5% of human serum albumin serum) (n=7) or (iii) placebo solution (1 mL saline solution with 2% of autologous serum) (n=10), which were administered into the periadventitial arteries.

The follow-up visits were at months 1, 3, 6, and 12, to evaluate the following parameters:

(i) Rutherford classification (0 to 6) (ii) TcPO2 (mmHg) (iii) Wound closure (area cm2) (iv) pain (visual analogue scale (0-10) (v) pain-free walking distance (m) (vi) revascularization and limb-survival proportion during follow-up (vii) the quality of life (EQ-5D questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 40 years of age or over (until 85 years old)
* TcPO2 ≤ 30 mmHg.
* Diagnosis of diabetes.
* Patients with signs of critical ischemia such as (i) ulcer that does not heal, (ii) necrosis or loss of tissue, (iii) pain at rest, and (iv) intermittent claudication.
* Basal Rutherford classification stage 3 to 5.
* Non-revascularizable patients due to comorbidities and/or anatomy.
* Patients that despite revascularization (vascular surgery), have adequate distal beds to perfuse the limb.
* Ankle/brachial index less than 0.4.
* Stenosis or occlusion of the infrapatellar arteries.

Exclusion Criteria:

* Participants that do not sign the informed consent.
* Presence of osteomyelitis.
* Hemodynamic instability (MAP<65 mmHg or vasopressor requirement).
* Any acute systemic infectious disease process.
* Severe sepsis.
* Uncontrolled coagulopathy.
* Condition of cancer.
* Use of immunosuppressive or cytotoxic drugs
* Alterations of the bone marrow that do not allow the adequate extraction of the components to be used as: acute leukemia, chronic leukemia, marrow aplasia, myelodysplastic syndrome, and myelophthisis.
* Contraindication of sedation for bone marrow aspirate.
* Patients who have suffered in a period < six months of myocardial infarction, disease cerebrovascular or coronary intervention.
* Patients with liver failure indicated by serum transaminases (aspartate aminotransferase and alanine aminotransferase), with values twice the normal limit.
* Any acute or chronic contagious disease including hepatitis B, hepatitis C, and HIV.
* Any other comorbidity that the treating vascular surgeon considers as a contraindication to cell treatments.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Safety profile: (adverse events (AEs) and serious AEs) | 12 months
  AEs: (i) local toxicity, including signs of local inflammation (swelling, warmth, impairment of function), worsening of ulcer, new ulcer, or hematomas after auto-BM-MNC or allo-WJ-MSCs administration.
  (ii) systemic toxicity as fever, allergies. (iii) maximum grade toxicity for tissue.
Safety profile | 12 months
  Serious AEs: hospitalization, malignancy, amputation, persistent or significant disability, or death.
Efficacy profile: Rutherford's classification | 12 months
  0 to 6
TcPO2 | 12 months
  mmHg
Efficacy profile: Visual Analogue Scale pain | 12 months
  0 to10
Efficacy profile: Pain-free walking distance | 12 months
  meters
Efficacy profile: Wound closure | 12 months
  cm2
Efficacy profile: Revascularization | 12 months
  Percentage
Efficacy profile: Limb survival proportion | 12 months
  Percentage
Efficacy profile: Quality of life | 12 months
  EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martha L Arango, PhD, Principal Investigator — Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Locations (1):
- Fundación Oftalmológica de Santander (FOSCAL), Bucaramanga, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arango-Rodriguez ML, Mateus LC, Sossa CL, Becerra-Bayona SM, Solarte-David VA, Ochoa Vera ME, Viviescas LTG, Berrio AMV, Serrano SE, Vargas O, Isla AC, Benitez A, Rangel G. A novel therapeutic management for diabetes patients with chronic limb-threatening ischemia: comparison of autologous bone marrow mononuclear cells versus allogenic Wharton jelly-derived mesenchymal stem cells. Stem Cell Res Ther. 2023 Aug 25;14(1):221. doi: 10.1186/s13287-023-03427-z. PMID 37626416